CLINICAL TRIAL: NCT04777890
Title: Effects of Instrumental, Manipulative and Soft Tissue Approaches for the Suboccipital Region in Subjects With Chronic Mechanical Neck Pain. A Randomized Controlled Trial
Brief Title: Effects of Instrumental and Manipulative Techniques for the Suboccipital Region in Subjects With Chronic Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Juan José Arjona Retamal (Other)
Responsible Party: Sponsor-Investigator, Juan José Arjona Retamal, Principal Investigator, Universidad Rey Juan Carlos
Organization: Universidad Rey Juan Carlos (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: University Rey Juan Carlos
Record Dates: First submitted 2021-02-20; First posted 2021-03-02 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Chronic Mechanical Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- suboccipital inhibition technique group (Active Comparator)
  Interventions: Other: suboccipital inhibition
- INYBI group (Experimental): Participants in this group will be treated with the INYBI, an instrument designed for treating the suboccipital area, in a more precise way than the manual technique.
  Interventions: Other: INYBI
- combined treatment group (Experimental): Participants in this group will be first treated with the INYBI and then receive an upper cervical manipulation
  Interventions: Other: INYBI + upper cervical manipulation

INTERVENTIONS:
Other: suboccipital inhibition — The therapist will seat at the patient's head height and place his second, third, fourth and fifth fingertips'over the patient's suboccipital area during a 10-minute period.
  Arms: suboccipital inhibition technique group
Other: INYBI — The therapist will place the INYBI at the suboccipital area, specifically placing the fingers of the instrument at the lower border of the occipital. If needed, a rolled towel will be placed behind the INYBI, in order to maintain the physiological lordosis, checking out that the patient doesn't make a cervical extension. Then the therapist will press the vibration button and turn it off after 10 minutes. All patients will receive the treatment with the INYBI's hardest head with a 50 HZ frequency.
  Arms: INYBI group
Other: INYBI + upper cervical manipulation — The participant will also be treated with the INYBI during a 10-minute period. After that, the therapist will carry out the upper cervical manipulation technique. Keeping the patient's head on an upper cervical flexion position, the therapist will turn his/her head to the maximum possible rotation, always maintaining its longitudinal axis. Once this is done, a high velocity and short articular amplitude manipulation in rotation will be carried out
  Arms: combined treatment group

SUMMARY:
The aim of the study is to compare the effectiveness between the suboccipital inhibition technique, the suboccipital inhibition carried out with the INYBI instrument and the suboccipital inhibition with the INYBI plus the upper cervical manipulation, all in patients with chronic mechanic cervicalgia, and to determine which of these techniques is the most effective in the variables studied. In order to do so, 96 subjects participated in the study, being assigned to the 3 intervention groups. We expected the combined treatment (INYBI instrument + upper cervical manipulation) to be the one to produce the best results.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged between 18 and 40 all diagnosed with chronic mechanic cervical pain with an evolution of at least 3 months and who show pain that increases with maintained postures, during movement and during spinal muscles palpation.

Exclusion Criteria:

* participants that can't read and/or fill in the informed consent, either due to a language and/or cognition alteration or age-related factors.
* subjects with psychological pathologies, such as hysteria, depression or anxiety.
* subjects that have received a manual treatment two months before the beginning of the clinical trial.
* subjects who have been recommended by a physician or an anesthetist to receive any type of analgesic, anti-inflammatory or neuromodulator medication, such as antidepressants, antiepileptics and benzodiazepines. If the patient took in this type of medication in an occasional way 72 hours before the beginning of the study, he/she could participate.
* the treatment and assessment techniques will be avoided if: fear to vertebral manipulation in the upper cervical area or positive Klein test and other integrity test of the vertebral artery, positive cervical instability test and positive Spurling test (foraminal compression test).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Changes in patients' cervical functionality between baseline and follow-up period. | Baseline and two weeks after the second intervention.
  cervical functionality is measured with the Neck Disability Index

SECONDARY OUTCOMES:
Changes in patients' cervical mobility between baseline and follow-up periods. | Baseline, 10 minutes after the first intervention, 1 week after the first intervention and 10 minutes after the second intervention.
  The movements that will be measured with the CROM® are: flexion, extension, right and left rotation, right and left side-bending.
Changes in patients' pressure pain threshold between baseline and follow-up periods. | Baseline, 10 minutes after the first intervention, 1 week after the first intervention and 10 minutes after the second intervention.
  The pressure pain threshold will be measured with an algometer (Mechanical Algometer Pain Test® de Wagner Instrument, USA) in the suboccipital and trapezius muscles (both left and right).
Changes in patients' pain due to movement between baseline and follow-up periods. | Baseline, 10 minutes after the first intervention, 1 week after the first intervention and 10 minutes after the second intervention.
  The movements that will be measured with the visual analogue scale (VAS) are: flexion, extension, right and left rotation, right and left side-bending.

CONTACTS AND LOCATIONS:
Locations (1):
- Ofistema, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berolo S, Wells RP, Amick BC 3rd. Musculoskeletal symptoms among mobile hand-held device users and their relationship to device use: A preliminary study in a Canadian university population. Appl Ergon. 2011 Jan;42(2):371-8. doi: 10.1016/j.apergo.2010.08.010. Epub 2010 Sep 15. PMID 20833387
- [Background] Cohen SP. Epidemiology, diagnosis, and treatment of neck pain. Mayo Clin Proc. 2015 Feb;90(2):284-99. doi: 10.1016/j.mayocp.2014.09.008. PMID 25659245
- [Background] Cote P, Cassidy DJ, Carroll LJ, Kristman V. The annual incidence and course of neck pain in the general population: a population-based cohort study. Pain. 2004 Dec;112(3):267-273. doi: 10.1016/j.pain.2004.09.004. PMID 15561381
- [Background] Dunning JR, Cleland JA, Waldrop MA, Arnot CF, Young IA, Turner M, Sigurdsson G. Upper cervical and upper thoracic thrust manipulation versus nonthrust mobilization in patients with mechanical neck pain: a multicenter randomized clinical trial. J Orthop Sports Phys Ther. 2012 Jan;42(1):5-18. doi: 10.2519/jospt.2012.3894. Epub 2011 Sep 30. PMID 21979312
- [Background] Dunning JR, Butts R, Mourad F, Young I, Fernandez-de-Las Penas C, Hagins M, Stanislawski T, Donley J, Buck D, Hooks TR, Cleland JA. Upper cervical and upper thoracic manipulation versus mobilization and exercise in patients with cervicogenic headache: a multi-center randomized clinical trial. BMC Musculoskelet Disord. 2016 Feb 6;17:64. doi: 10.1186/s12891-016-0912-3. PMID 26852024
- [Background] Espi-Lopez GV, Gomez-Conesa A, Gomez AA, Martinez JB, Pascual-Vaca AO, Blanco CR. Treatment of tension-type headache with articulatory and suboccipital soft tissue therapy: A double-blind, randomized, placebo-controlled clinical trial. J Bodyw Mov Ther. 2014 Oct;18(4):576-85. doi: 10.1016/j.jbmt.2014.01.001. Epub 2014 Jan 10. PMID 25440210
- [Background] Espi-Lopez GV, Zurriaga-Llorens R, Monzani L, Falla D. The effect of manipulation plus massage therapy versus massage therapy alone in people with tension-type headache. A randomized controlled clinical trial. Eur J Phys Rehabil Med. 2016 Oct;52(5):606-617. Epub 2016 Mar 18. PMID 26989818
- [Background] Field, A. Discovering statistics using IBM SPSS statistics. Fourth Edition. London. Sage; 2013. pp. 473-474.
- [Background] Galindez-Ibarbengoetxea X, Setuain I, Ramirez-Velez R, Andersen LL, Gonzalez-Izal M, Jauregi A, Izquierdo M. Short-term effects of manipulative treatment versus a therapeutic home exercise protocol for chronic cervical pain: A randomized clinical trial. J Back Musculoskelet Rehabil. 2018 Feb 6;31(1):133-145. doi: 10.3233/BMR-169723. PMID 28826170
- [Background] Hoy D, March L, Woolf A, Blyth F, Brooks P, Smith E, Vos T, Barendregt J, Blore J, Murray C, Burstein R, Buchbinder R. The global burden of neck pain: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1309-15. doi: 10.1136/annrheumdis-2013-204431. Epub 2014 Jan 30. PMID 24482302
- [Background] Jimenez-Sanchez S, Fernandez-de-Las-Penas C, Carrasco-Garrido P, Hernandez-Barrera V, Alonso-Blanco C, Palacios-Cena D, Jimenez-Garcia R. Prevalence of chronic head, neck and low back pain and associated factors in women residing in the Autonomous Region of Madrid (Spain). Gac Sanit. 2012 Nov-Dec;26(6):534-40. doi: 10.1016/j.gaceta.2011.10.012. Epub 2012 Feb 18. PMID 22342049
- [Background] Jussila L, Paananen M, Nayha S, Taimela S, Tammelin T, Auvinen J, Karppinen J. Psychosocial and lifestyle correlates of musculoskeletal pain patterns in adolescence: a 2-year follow-up study. Eur J Pain. 2014 Jan;18(1):139-46. doi: 10.1002/j.1532-2149.2013.00353.x. Epub 2013 Jul 12. PMID 23853106
- [Background] Lee SP, Hsu YT, Bair B, Toberman M, Chien LC. Gender and posture are significant risk factors to musculoskeletal symptoms during touchscreen tablet computer use. J Phys Ther Sci. 2018 Jun;30(6):855-861. doi: 10.1589/jpts.30.855. Epub 2018 Jun 12. PMID 29950780
- [Background] Medina i Mirapeix, F., Mantilla-Herrador, J. and Meseguer-Henajeros, A.B. (2000): "Guía de práctica clínica para el tratamiento y seguimiento fisioterápico de la cervicalgia mecánica", Fisioterapia, 22(S2), pp. 33-46.
- [Background] Namwongsa S, Puntumetakul R, Neubert MS, Boucaut R. Factors associated with neck disorders among university student smartphone users. Work. 2018;61(3):367-378. doi: 10.3233/WOR-182819. PMID 30373996
- [Background] Nestares MT, Salinas M, De Teresa C, Diaz-Castro J, Moreno-Fernandez J, Lopez-Frias M. [Risk factors related with lifestyle in patients with musculoskeletal disorders]. Nutr Hosp. 2017 Mar 30;34(2):444-453. doi: 10.20960/nh.237. Spanish. PMID 28421803
- [Background] Prushansky T, Dvir Z, Defrin-Assa R. Reproducibility indices applied to cervical pressure pain threshold measurements in healthy subjects. Clin J Pain. 2004 Sep-Oct;20(5):341-7. doi: 10.1097/00002508-200409000-00009. PMID 15322441
- [Background] Shan Z, Deng G, Li J, Li Y, Zhang Y, Zhao Q. Correlational analysis of neck/shoulder pain and low back pain with the use of digital products, physical activity and psychological status among adolescents in Shanghai. PLoS One. 2013 Oct 11;8(10):e78109. doi: 10.1371/journal.pone.0078109. eCollection 2013. PMID 24147114
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543
- [Background] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753
- [Background] Vernon H. The Neck Disability Index: state-of-the-art, 1991-2008. J Manipulative Physiol Ther. 2008 Sep;31(7):491-502. doi: 10.1016/j.jmpt.2008.08.006. PMID 18803999
- [Background] Waalen, D., White, P. and Waalen, J. (1994): "Demographic and clinical characteristics of chiropractic patients: A 5-year study of patients trated at the Canadian Memorial Chiropractic College", The journal of the CCA, 38(2), pp. 75-82.
- [Background] Xie Y, Szeto GP, Dai J, Madeleine P. A comparison of muscle activity in using touchscreen smartphone among young people with and without chronic neck-shoulder pain. Ergonomics. 2016;59(1):61-72. doi: 10.1080/00140139.2015.1056237. Epub 2015 Jul 28. PMID 26218600
- [Background] Perez-Martinez C, Gogorza-Arroitaonandia K, Heredia-Rizo AM, Salas-Gonzalez J, Oliva-Pascual-Vaca A. INYBI: A New Tool for Self-Myofascial Release of the Suboccipital Muscles in Patients With Chronic Non-Specific Neck Pain: A Randomized Controlled Trial. Spine (Phila Pa 1976). 2020 Nov 1;45(21):E1367-E1375. doi: 10.1097/BRS.0000000000003605. PMID 32796456